CLINICAL TRIAL: NCT02655146
Title: Implantation in Frozen Embryo Transfer
Brief Title: the Effects of GnRHa Add up to Routine Luteal Phase Support on Frozen Embryo Implantation in Frozen Embryo Transfer .
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Qing Reproducive and Genetic Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ferring-IIT-01
Record Dates: First submitted 2016-01-12; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
Keywords: Frozen embryo transfer,luteal support, GnRHa
MeSH Terms: conditions — Infertility | interventions — Estradiol; Progesterone; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GnRHa protocol (Experimental): All subjects are artificially preparing endometrium starting on day 3-5 of the cycle with oral E2 (Progynova) 4-10mg/day at least 14 days. After ultrasound and hormone tests, progesterone 100mg/day intramuscular injection is allocated with E2.In the meanwhile, if the subjects have a fail history of hormonal artificially preparing endometrium, such as an early ovulation, a singal dose of triptorelin 3.75mg would be intramuscular injected before E2 was used as a pretreatment. Then a maximum of two embryos are transferred when endometrium is perfectly prepared. All subjects receive routine luteal phase support with E2 and progesterone .A single dose of Triptorelin 0.1mg is administrated on the 3rd day after embryo implanted with routine luteal phase support.
  Interventions: Drug: triptorelin 0.1; Drug: E2; Drug: Progesterone; Drug: triptorelin 3.75mg
- routine luteal phase protocol (Other): All subjects are artificially preparing endometrium starting on day 3-5 of the cycle with oral E2 4-10mg/day at least 14 days. After ultrasound and hormone tests, progesterone 100mg/day intramuscular injection is allocated with E2. In the meanwhile, if the subjects have a fail history of hormonal artificially preparing endometrium, such as an early ovulation, a singal dose of triptorelin 3.75mg would be intramuscular injected before E2 was used as a pretreatment. Then a maximum of two embryos are transferred when endometrium is perfectly prepared. All subjects receive routine luteal phase support with E2 and progesterone .
  Interventions: Drug: E2; Drug: Progesterone; Drug: triptorelin 3.75mg

INTERVENTIONS:
Drug: triptorelin 0.1 — a single dose of decapeptyl 0.1 s.c. on the 3rd day of embryo transfer with routine luteal phase support.
  Other Names: decapeptyl 0.1
  Arms: GnRHa protocol
Drug: E2 — Patients will be on the Progynova tablets 4-10mg daily at least 14 days.
  Other Names: Progynova
Drug: Progesterone — After ultrasound and hormorne tests, progesterone 100mg intramuscular injection is allocated with Progynova.
Drug: triptorelin 3.75mg — as a pretreatment of E2 in some subjects with a fail history of hormonal artificially endometrium preparing.
  Other Names: Diphereline 3.75mg

SUMMARY:
The aim of the present prospective randomized controlled study was to determine the effects of GnRHa add up to routine luteal phase support on frozen embryo implantation in frozen embryo transfer (FET).

DETAILED DESCRIPTION:
Some recent data have suggested a beneficial effect of GnRHa administered in the luteal phase on the outcome of assisted reproduction techniques. In those studies, the dose and administration time of GnRHa are inconsistent. Single administration on third day after embryo transfer and multiple dose injection during luteal phase are the most common way. The GnRHa included Triptorelin 0.1mg, Leuprorelin 1mg and Buserelin 600ug et al. The exact underlying mechanism is still not clear, although it has been hypothesized that GnRH agonist either supports the corpus luteum function by inducing LH secretion by the pituitary gonadotrophin cells or stimulates the endometrium GnRH receptors . Tesarik et al.postulated a direct effect of GnRH agonist on the embryo, evidenced by increased β-HCG secretion.

Currently, available data suggest that inadvertent administration of a GnRH agonist during a conception cycle is not accompanied by an increased risk of birth defects. On the basis of the currently strong available evidence, it appears that GnRH agonist supplementation during luteal phase significantly improve the outcome of ART treatment. Most of the former researches focused only on fresh embryo transfer in IVF/ICSI cycles. In one prospective controlled study, a single dose of Triptorelin 0.1mg was administrated 6 days after ICSI in oocyte donor cycles and the implantation rate was improved significantly.GnRH agonist administration at the time of implantation enhances embryo developmental potential, probably by a direct effect on the embryo.

ELIGIBILITY:
Inclusion Criteria:

* infertile women with frozen thawed embryo transfer after HRT endometrial preparation.
* more than 20 years old, and less than 37 years old.
* BMI less than 28kg/m2.
* more than 1 transplantable embryo after thawing.
* patients should sign the informed consent and have the willing to follow up.

Exclusion Criteria:

* uterine malformation
* diameter of intramural myoma more than 3cm
* the thickness of endometrium less than 7mm on the progesterone supportive day.

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
implantation rate | 5 weeks

SECONDARY OUTCOMES:
clinical pregancy rate | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ye, bachelor, Study Director — chong qing reproductive and genetic institute
Locations (1):
- Chong Qing Reproductive and Genetic Institute, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Linden M, Buckingham K, Farquhar C, Kremer JA, Metwally M. Luteal phase support for assisted reproduction cycles. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD009154. doi: 10.1002/14651858.CD009154.pub2. PMID 21975790